CLINICAL TRIAL: NCT02027571
Title: Pathobiology and Reversibility of Prediabetes in a Biracial Cohort (PROP-ABC)
Brief Title: Pathobiology and Reversibility of Prediabetes in a Biracial Cohort
Acronym: PROP-ABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB Number: 12-01970-FB; R01DK067269 (NIH)
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2016-10

CONDITIONS: Prediabetes; Type 2 Diabetes; Obesity
Keywords: Diabetes; Race/Ethnicity; Offspring Cohort; African Americans; Prediabetes Reversal; Lifestyle Intervention; Insulin Sensitivity; Beta-cell Function; Diabetes Prevention
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensive Lifestyle Intervention (ILI) (Experimental): ILI consists of weight loss ( > 10%); caloric reduction; physical activity (180 min/week); monthly visits for group counseling for 6 months, followed by quarterly visits; and meal replacements.
  Interventions: Behavioral: Intensive Lifestyle Intervention (ILI)

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention (ILI) — ILI consists of weight loss ( > 10%); caloric reduction; physical activity (180 min/week); monthly visits for group counseling for 6 months, followed by quarterly visits; and meal replacements.

SUMMARY:
The reasons for the epidemics of diabetes and prediabetes, and why individuals from certain populations suffer at higher rates are not well known. In the Pathobiology and Reversibility of Prediabetes in a Biracial Cohort (PROP-ABC) study, nearly 400 African Americans and Caucasians whose parents have type 2 diabetes will undergo repeated testing to determine what factors lead to the occurrence of prediabetes, and whether race still plays a major role in a setting where everyone being studied has one or both parents with diabetes. The PROP-ABC Study also will test the hypothesis that the ability of intensive lifestyle intervention to reverse prediabetes and return people's metabolism back to normal is dependent on how long people have had prediabetes.

DETAILED DESCRIPTION:
The Pathobiology and Reversibility of Prediabetes in a Biracial Cohort (PROP-ABC) study is following an extant cohort of 376 initially normoglycemic African American and Caucasian offspring of parents with type 2 diabetes for an additional 5years. The subjects were enrolled between 2006 and 2009 and have been followed up to 2012, during which 10 have developed diabetes and 101 developed prediabetes, without evidence of racial disparities.

The objectives of PROP-ABC are to gain a fuller understanding of the natural history and predictors of early glucose abnormalities, determine the role of race during the second wave of glycemic progression, and to access the time dependency of reversibility of prediabetes. The study tests 4 hypotheses: 1) Among offspring of parents with type 2 diabetes, early progression from normal to impaired glucose regulation (within 5 yr) occurs in the highest-risk subjects independently of race, whereas late progression (5-10 yr) displays racial disparities, and is predicted by physiological, biochemical and behavioral markers; 2) Early microvascular complications, peripheral vascular disease (PVD), and endothelial dysfunction manifest during transition from normal to impaired glucose regulation, display racial disparities, and are predicted by glycemic and nonglycemic factors; 3) The "metabolically healthy" insulin-sensitive obese (ISO) phenotype displays racial disparities in its association with cardiometabolic risk factors and incident dysglycemia among African-Americans and Caucasians offspring of parents with type 2 diabetes; and 4) Duration of the prediabetic state is a major determinant of, and is inversely related to, the efficacy of lifestyle intervention to induce regression of the prediabetic phenotype and restoration of normal glucose regulation. Participants with prediabetes and others who develop prediabetes during PROP-ABC will receive Intensive Lifestyle intervention (ILI).

We define duration of prediabetes as the interval from date of confirmed prediabetes to the date of initiation of ILI, stratified to 3 prediabetes intervals: a) <1 yr, b) 1 to <3 yr, c) 3-6 yr. The primary outcome measure is restoration of normal glucose regulation (fasting plasma glucose <100 mg/dl and 2-hour post-load plasma glucose < 140 mg/dl). Secondary endpoints include normalization of either fasting plasma glucose or 2-hour post-load plasma glucose , occurrence of diabetes, insulin sensitivity and secretion. Data will be analyzed according to the "intention to treat" principle. Based on power calculations, a sample size of 150 subjects (50/prediabetes interval) would allow detection of medium to large effect off ILI with ~85% power. Kaplan-Meier survival curves will be generated for the 3 prediabetes intervals, and log-rank test will be used to analyze the time to occurrence of primary outcome. The prospective PROP-ABC, designed to identify new cases of prediabetes as they occur, is uniquely placed to test the time dependency of reversibility of incident prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* As planned these studies will enroll interested persons from among the group of 376 subjects who participated in the Pathobiology of Prediabetes in a Biracial Cohort (POP-ABC) study between 2006 and 2012. That group includes 267 women and 109 men; 217 are African Americans and 159 are Caucasians. At the time of initial enrollment into POP-ABC, these participants were selected for being nondiabetic offspring of parents with type 2 diabetes. Race and ethnicity was by self-report of non-Hispanic white or non-Hispanic black heritage, and their age range was 18-65 years at enrollment. No new subjects will be recruited into this established cohort. To be eligible for inclusion in the renewal study, subjects must be ambulatory, be in good general health, and must not be taking medications known to alter insulin sensitivity, insulin secretion, or body weight.

Exclusion Criteria:

* Exclusion criteria: Persons not enrolled in POP-ABC study; diagnosis of diabetes or use of any antidiabetic medication; medical conditions that preclude participation in physical activity; history of liposuction, surgical weight reduction; use of glucocorticoids, beta-blockers, thiazide diuretics (> 25 mg/day), or medication known to alter glucose metabolism. Women who are pregnant or become pregnant while participating in this study will have all testing procedures delayed until 12 months after delivery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is restoration of normal glucose regulation | Up to 60 months
  The primary outcome measure is restoration of normal glucose regulation (FPG <100 mg/dl and 2hrPG < 140 mg/dl).

SECONDARY OUTCOMES:
Glucose normalization | Up to 60 months
  Secondary endpoints include normalization of either fasting plasma glucose or 2-hr OGTT plasma glucose levels, occurrence of diabetes, insulin sensitivity and secretion.

OTHER OUTCOMES:
Incident prediabetes in observational cohort | Up to 60 months
  Incident prediabetes, microvascular complications, endothelial function, ankle-brachial index, body composition, adiposity measures, FPG, 2hPG , A1c, adipo- and inflammatory cytokines (hsCRP, TNF-a, IL-1a, IL-6, resistin, leptin and adiponectin), metabolic syndrome and individual components (waist, BP, triglycerides, HDL cholesterol, FPG), metabolically healthy and unhealthy obese phenotypes, transaminases (surrogate for liver fat), diet (FHQ score) physical activity (MAQ and NHANES scores) and smoking history.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Dagogo-Jack, MD, Principal Investigator — University of Tennessee
Locations (1):
- Clinical Research Center, University of Tennessee Health Scienc Ctr, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Group data will be published after completion of study and analysis of results. Individual participant-level information will not be shared.

REFERENCES:
- [Background] Dagogo-Jack S, Edeoga C, Ebenibo S, Chapp-Jumbo E; Pathobiology of Prediabetes in a Biracial Cohort (POP-ABC) Research Group. Pathobiology of Prediabetes in a Biracial Cohort (POP-ABC) study: baseline characteristics of enrolled subjects. J Clin Endocrinol Metab. 2013 Jan;98(1):120-8. doi: 10.1210/jc.2012-2902. Epub 2012 Nov 1. PMID 23118422
- [Background] Ebenibo S, Edeoga C, Ammons A, Egbuonu N, Dagogo-Jack S; Pathobiology of Prediabetes in a Biracial Cohort (POP-ABC) Research Group. Recruitment strategies and yields for the Pathobiology of Prediabetes in a Biracial Cohort: a prospective natural history study of incident dysglycemia. BMC Med Res Methodol. 2013 May 10;13:64. doi: 10.1186/1471-2288-13-64. PMID 23663750
- [Background] Dagogo-Jack S, Edeoga C, Ebenibo S, Nyenwe E, Wan J; Pathobiology of Prediabetes in a Biracial Cohort (POP-ABC) Research Group. Lack of racial disparity in incident prediabetes and glycemic progression among black and white offspring of parents with type 2 diabetes: the pathobiology of prediabetes in a biracial cohort (POP-ABC) study. J Clin Endocrinol Metab. 2014 Jun;99(6):E1078-87. doi: 10.1210/jc.2014-1077. Epub 2014 Mar 14. PMID 24628558
- [Background] Owei I, Umekwe N, Wan J, Dagogo-Jack S. Plasma lipid levels predict dysglycemia in a biracial cohort of nondiabetic subjects: Potential mechanisms. Exp Biol Med (Maywood). 2016 Nov;241(17):1961-1967. doi: 10.1177/1535370216659946. Epub 2016 Jul 17. PMID 27430991
- [Background] Nyenwe E, Owei I, Wan J, Dagogo-Jack S. Parental History of Type 2 Diabetes Abrogates Ethnic Disparities in Key Glucoregulatory Indices. J Clin Endocrinol Metab. 2018 Feb 1;103(2):514-522. doi: 10.1210/jc.2017-01895. PMID 29216357
- [Background] Edeoga C, Owei I, Siwakoti K, Umekwe N, Ceesay F, Wan J, Dagogo-Jack S. Relationships between blood pressure and blood glucose among offspring of parents with type 2 diabetes: Prediction of incident dysglycemia in a biracial cohort. J Diabetes Complications. 2017 Nov;31(11):1580-1586. doi: 10.1016/j.jdiacomp.2017.07.019. Epub 2017 Aug 2. PMID 28890305
- [Result] Owei I, Umekwe N, Mohamed H, Ebenibo S, Wan J, Dagogo-Jack S. Ethnic Disparities in Endothelial Function and Its Cardiometabolic Correlates: The Pathobiology of Prediabetes in A Biracial Cohort Study. Front Endocrinol (Lausanne). 2018 Mar 13;9:94. doi: 10.3389/fendo.2018.00094. eCollection 2018. PMID 29593654
- [Result] Owei I, Umekwe N, Provo C, Wan J, Dagogo-Jack S. Insulin-sensitive and insulin-resistant obese and non-obese phenotypes: role in prediction of incident pre-diabetes in a longitudinal biracial cohort. BMJ Open Diabetes Res Care. 2017 Jul 19;5(1):e000415. doi: 10.1136/bmjdrc-2017-000415. eCollection 2017. PMID 28878939
- [Derived] Dagogo-Jack S, Umekwe N, Brewer AA, Owei I, Mupparaju V, Rosenthal R, Wan J. Outcome of lifestyle intervention in relation to duration of pre-diabetes: the Pathobiology and Reversibility of Prediabetes in a Biracial Cohort (PROP-ABC) study. BMJ Open Diabetes Res Care. 2022 Mar;10(2):e002748. doi: 10.1136/bmjdrc-2021-002748. PMID 35273012
- [Derived] Dagogo-Jack S, Brewer AA, Owei I, French L, Umekwe N, Rosenthal R, Wan J. Pathobiology and Reversibility of Prediabetes in a Biracial Cohort (PROP-ABC) Study: design of lifestyle intervention. BMJ Open Diabetes Res Care. 2020 Jun;8(1):e000899. doi: 10.1136/bmjdrc-2019-000899. PMID 32527719